CLINICAL TRIAL: NCT02159352
Title: A Phase 1 Clinical Study to Assess the Effect of Darunavir/Ritonavir or Lopinavir/Ritonavir on the Pharmacokinetics of Daclatasvir in Healthy Subjects
Brief Title: Study Assessing the Effects of Darunavir/Ritonavir or Lopinavir/Ritonavir on the Pharmacokinetics of Daclatasvir in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AI444-093
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Darunavir; Ritonavir; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Daclatasvir and Darunavir/Ritonavir (Experimental): Treatment A: Daclatasvir oral tablet on specific days
  Treatment B: Daclatasvir tablet and Darunavir Tablet/Ritonavir capsule orally on specific days
  Interventions: Drug: Daclatasvir; Drug: Darunavir; Drug: Ritonavir
- Group 2: Daclatasvir and Lopinavir/Ritonavir (Experimental): Treatment C: Daclatasvir oral tablet on specific days
  Treatment D: Daclatasvir tablet and Lopinavir/Ritonavir tablet orally on specific days
  Interventions: Drug: Daclatasvir; Drug: Ritonavir; Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Daclatasvir
  Other Names: BMS-790052
Drug: Darunavir
  Other Names: Prezista
  Arms: Group 1: Daclatasvir and Darunavir/Ritonavir
Drug: Ritonavir
  Other Names: Norvir
Drug: Lopinavir/Ritonavir
  Arms: Group 2: Daclatasvir and Lopinavir/Ritonavir

SUMMARY:
The purpose of this study is to determine whether multiple doses of darunavir/ritonavir or lopinavir/ritonavir affect the pharmacokinetics of daclatasvir in healthy participants.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Healthy male and female participants, aged 18 to 49, as determined by medical history, physical examination, 12 lead electrocardiogram, vital signs, and clinical laboratory evaluations

Key Exclusion Criteria:

* Any significant acute or chronic medical illness; donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration (within 2 weeks for plasma only); or blood screen findings positive for hepatitis C antibody, hepatitis B surface antigen, or HIV-1 and HIV-2 antibodies

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Healthcare Discoveries, Llc D/B/A Icon Development Solutions, San Antonio, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 site in the United States of America.
Pre-assignment Details: Of 49 participants enrolled, 28 were randomized to receive treatment. Of the 21 who were not randomized, 16 no longer met study criteria and 5 discontinued due to other reasons.
Groups:
- Daclatasvir + Darunavir/Ritonavir: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4 and a 30-mg daclatasvir tablet once daily, along with an 800-mg darunavir tablet and a 100-mg ritonavir capsule once daily on Days 5 through 14.
- Daclatasvir + Lopinavir/Ritonavir: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4 and a 30-mg daclatasvir tablet once daily, along with 2 200-mg lopinavir/50-mg ritonavir tablets twice daily on Days 5 through 14.
Period: Overall Study
Arm/Group | Daclatasvir + Darunavir/Ritonavir | Daclatasvir + Lopinavir/Ritonavir
Started | 14 | 14
Phase 1 (Day 1- 4) | 14 | 14
Phase 2 (Day 5-14) | 11 | 12
Completed | 11 | 12
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daclatasvir + Darunavir/Ritonavir | Daclatasvir + Lopinavir/Ritonavir | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Daclatasvir
Description: Cmax was obtained from concentration-time plot using a noncompartmental method and a validated pharmacokinetic analysis program.
Time Frame: Predose (0 hour) on Day 2, 3 and 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hours on Day 4 (Period 1); Predose (0 hour) on Day 12, 13 and 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 hour on Day 14 (Period 2)
Population: All treated participants with adequate pharmacokinetic profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 1: Daclatasvir (60 mg): Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4.
- Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily, along with an 800-mg darunavir tablet, and a 100-mg ritonavir capsule once daily on Days 5 through 14.
- Group 2: Daclatasvir (60 mg): Participants received a 60-mg daclatasvir tablet once daily on Days 5 through 14.
- Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with 2 200-mg lopinavir/50-mg ritonavir tablets twice daily Days 5 through 14.
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 11 | 14 | 13
ng/mL | 1335 (38) | 493 (36) | 1412 (28) | 476 (21)
Statistical Analysis 1: Comparison: Group 1: Daclatasvir (60 mg) vs Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir; A general linear mixed effect model (restricted maximum likelihood) with treatment as fixed effect and measurements within each participant as repeated measures was fitted to the log-transformed Cmax; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 0.384, 90% CI 2-sided [0.348 to 0.423]
Statistical Analysis 2: Comparison: Group 2: Daclatasvir (60 mg) vs Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 0.337, 90% CI 2-sided [0.306 to 0.371]

2. Primary Outcome: Area Under the Concentration-Time Curve in 1 Dosing Interval (AUC[TAU]) for Daclatasvir
Description: AUC(TAU) was the area under the curve from time zero to end of dosing interval. AUC(TAU) was obtained from concentration-time plot of daclatasvir using noncompartmental method and a validated pharmacokinetic analysis program.
Time Frame: as for outcome 1
Population: All treated participants with adequate pharmacokinetic profiles. Number of participants analyzed (N) signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Daclatasvir (60 mg) Days 1-4: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4.
- Daclatasvir (30 mg) + Darunavir/Ritonavir Days 5-14: Participants received a 30-mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and a 100-mg ritonavir capsule once daily on Days 5 through 14.
- Daclatasvir (60 mg) Days 5-14: Participants received a 60-mg daclatasvir tablet once daily on Days 5 through 14.
- Daclatasvir (30 mg) + Lopinavir/Ritonavir Days 5-14: Participants received a 30-mg daclatasvir tablet once daily along with 2 200-mg lopinavir/50-mg ritonavir tablets twice daily Days 5 through 14.
Arm/Group | Daclatasvir (60 mg) Days 1-4 | Daclatasvir (30 mg) + Darunavir/Ritonavir Days 5-14 | Daclatasvir (60 mg) Days 5-14 | Daclatasvir (30 mg) + Lopinavir/Ritonavir Days 5-14
Number analyzed (Participants) | 14 | 11 | 14 | 12
ng*h/mL | 12677 (41) | 8295 (39) | 13799 (26) | 7855 (23)
Statistical Analysis 1: Comparison: Daclatasvir (60 mg) Days 1-4 vs Daclatasvir (30 mg) + Darunavir/Ritonavir Days 5-14; A general linear mixed effect model (restricted maximum likelihood) with treatment as fixed effect and measurements within each participant as repeated measures was fitted to the log-transformed AUC(TAU); Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 0.703, 90% CI 2-sided [0.658 to 0.750]
Statistical Analysis 2: Comparison: Daclatasvir (60 mg) Days 5-14 vs Daclatasvir (30 mg) + Lopinavir/Ritonavir Days 5-14; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 0.577, 90% CI 2-sided [0.535 to 0.622]

3. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Daclatasvir
Description: Tmax was obtained from concentration-time plot of daclatasvir by using non-compartmental method by a validated pharmacokinetic analysis program.
Time Frame: as for outcome 1
Population: All treated participants with adequate pharmacokinetic profile. Here, N signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: hours
Groups:
- Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and a 100-mg ritonavir capsule once daily on Days 5 through 14.
- Group 2: Daclatasvir (60 mg): Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4.
- Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with 2 200-mg lopinavir/50-mg ritonavir tablets twice daily on Days 5 through 14.
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 11 | 14 | 13
hours | 2.00 [1.00 to 6.00] | 3.00 [1.00 to 6.00] | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 11.93]

4. Secondary Outcome: Plasma Concentration Observed at 24 Hours Postdose (C24) of Daclatasvir
Description: C24 was obtained from concentration time plot of daclatasvir by using noncompartmental method by a validated pharmacokinetic analysis program.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Group 2: Daclatasvir (60 mg): Participants received 60 mg of daclatasvir tablet once daily from Day 1 through 4.
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 11 | 14 | 12
ng/mL | 225 (54) | 250 (45) | 225 (36) | 280 (29)

5. Secondary Outcome: Dose-normalized Maximum Observed Plasma Concentration (Cmax/D) and Dose-normalized Plasma Concentration Observed at 24 Hours Postdose (C24/D) of Daclatasvir
Description: Cmax/D and C24/D are obtained from concentration-time plot of daclatasvir by using noncompartmental method by a validated pharmacokinetic analysis program.
Time Frame: as for outcome 1
Population: All treated participants with adequate pharmacokinetic profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Groups:
- Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with 2 200-mg lopinavir/ 50-mg ritonavir tablets twice daily on Days 5 through 14.
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 11 | 14 | 13
ng/mL/mg
  Cmax/D | 22.2 (38) | 16.4 (36) | 23.5 (28) | 15.9 (21)
  C24/D | 3.75 (54) | 8.34 (45) | 3.76 (36) | 9.33 (29)
Statistical Analysis 1: Comparison: Group 1: Daclatasvir (60 mg) vs Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir; A general linear mixed effect model (restricted maximum likelihood) with treatment as fixed effect and measurements within each participant as repeated measures was fitted to the log-transformed Cmax/D; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 0.768, 90% CI 2-sided [0.697 to 0.846]
Statistical Analysis 2: Comparison: Group 2: Daclatasvir (60 mg) vs Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 0.673, 90% CI 2-sided [0.611 to 0.742]

6. Secondary Outcome: Dose-normalized Area Under the Concentration-Time Curve in 1 Dosing Interval (AUC[TAU]/D) of Daclatasvir
Description: AUC(TAU)/D was obtained from concentration-time plot of daclatasvir by using noncompartmental method by a validated pharmacokinetic analysis program.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h/mL)/mg
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 11 | 14 | 12
(ng*h/mL)/mg | 211 (41) | 276 (39) | 230 (26) | 262 (23)
Statistical Analysis 1: Comparison: Group 1: Daclatasvir (60 mg) vs Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir; A general linear mixed effect model (restricted maximum likelihood) with treatment as fixed effect and measurements within each participant as repeated measures was fitted to the log-transformed (AUC(TAU)/D); Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 1.406, 90% CI 2-sided [1.317 to 1.501]
Statistical Analysis 2: Comparison: Group 2: Daclatasvir (60 mg) vs Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Adjusted Geometric Mean Ratio = 1.154, 90% CI 2-sided [1.070 to 1.244]

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Discontinuations Due to Adverse Events (AEs) and Who Died
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization.
Time Frame: From start of study treatment (Day 1) to study discharge for AEs (up to 15 days); Day 1 to 30 days after last dose of study treatment for SAEs (up to 44 days)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with 2 -mg lopinavir/50-mg ritonavir tablets twice daily on Days 5 through 14.
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants
  SAE | 0 | 0 | 0 | 0
  Discontinued due to AEs | 0 | 3 | 0 | 1
  Death | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormalities in Vital Sign Measurements
Description: Criteria for abnormalities in vital sign measurements: Diastolic blood pressure: Value >90 and change from baseline > 0 or value < 55 and change from baseline <-10. Systolic blood pressure: Value >140 and change from baseline >20 or value <90 and change from baseline <-20. Heart rate: Value >100 and change from baseline >30 or value <55 and change from baseline <-15. Respiration: Value >16 or change from baseline >10. Temperature: Value >38.3°C or change from baseline >1.6°C.
Time Frame: From start of study treatment (Day 1) to study discharge (up to 15 days)
Population: Participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Group 1: Daclatasvir + Darunavir/Ritonavir: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4 and a 30-mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and a 100-mg ritonavir capsule once daily on Days 5 through 14.
- Group 2: Daclatasvir + Lopinavir/Ritonavir: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4 and a 30-mg daclatasvir tablet once daily, along with 2 200-mg lopinavir/50-mg ritonavir tablets twice daily on Days 5 through 14.
Arm/Group | Group 1: Daclatasvir + Darunavir/Ritonavir | Group 2: Daclatasvir + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 14
participants | 3 | 2

9. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiogram (ECG) Findings
Description: Abnormalities in ECG findings included: PR ≥210 msec, QRS ≥120 msec, QT ≥500 msec, QTcF ≥450 msec, and second- or third-degree heart block.
Time Frame: From start of study treatment (Day 1) to study discharge (up to 15 days)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and 100-mg ritonavir capsule once daily on Days 5 through 14.
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants
  PR >210 | 2 | 4 | 0 | 1
  QRS >120 | 0 | 0 | 0 | 0
  QT >500 | 0 | 0 | 0 | 0
  QTcF >450 | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With Marked Abnormalities in Hematology Laboratory Test Results
Description: Criteria for marked abnormalities in test results: Platelet count >1.5*upper limits of normal (ULN) value, >1.5*ULN if pretreatment (PreRx) value is missing, <0.85*lower limit of normal (LLN) if PreRx ≥LLN, <0.85*LLN if PreRx is missing, <0.85*PreRx if PreRx <LLN. Leukocytes >1.2*ULN if LLN ≤PreRx ≤ULN, >1.2*ULN if PreRx is missing, >1.5*PreRx if PreRx >ULN, >ULN if PreRx <LLN, <0.85*PreRx if PreRx <LLN, <0.9*LLN if LLN ≤PreRx ≤ULN, <0.9*LLN if PreRx is missing and <LLN if PreRx >ULN. Lymphocytes >7.5*10^3 c/uL and <0.75*10^3 c/uL. Neutrophils <0.85*PreRx if PreRx <1.5*ULN, <1.5*ULN if PreRx ≥1.5*ULN and <1.5*ULN if PreRx is missing.
Time Frame: From start of study treatment (Day 1) to study discharge (up to 15 days)
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants
  Platelet Count | 1 | 0 | 0 | 0
  Leukocytes | 0 | 1 | 1 | 1
  Neutrophils (absolute) | 0 | 2 | 1 | 0
  Lymphocytes (absolute) | 0 | 1 | 0 | 0

11. Secondary Outcome: Number of Participants With Abnormalities in Urinalysis and Other Chemistry Testing Results
Description: Criteria for marked abnormalities on laboratory test results: urinary dipstick blood: ≥2 if pretreatment (PreRx) <1, ≥2 if PreRx is missing or ≥2*PreRx if PreRx ≥1. Urinary microscopic red blood cell (RBC): ≥2 if PreRx <2, ≥2 if PreRx is missing or ≥4 if PreRx ≥2. Urinary microscopic white blood cell (WBC): ≥2 if PreRx <2, ≥2 if PreRx is missing or ≥4 if PreRx ≥2. Lactate dehydrogenase >1.25*upper limit of normal (ULN) if PreRx ≤ULN, >1.25*ULN if PreRx is missing and >1.5*PreRx if PreRx >ULN.
Time Frame: From start of study treatment (Day 1) to study discharge (up to 15 days)
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Number analyzed (Participants) | 14 | 14 | 14 | 14
participants
  Blood, urine | 2 | 1 | 1 | 0
  RBC, urine | 1 | 1 | 0 | 0
  WBC, urine | 1 | 3 | 0 | 0
  Lactate dehydrogenase | 2 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: From start of study treatment (Day 1) to study discharge for AEs (up to 15 days); Day 1 to 30 days after last dose of study treatment for SAEs (up to 44 days)
Groups:
- Group 1: Total: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4 and 30 mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and a 100-mg of ritonavir capsule once daily on Days 5 through 14.
- Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir: Participants received a 30-mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and a 100-mg of ritonavir capsule once daily on Days 5 through 14.
- Group 2: Total: Participants received a 60-mg daclatasvir tablet once daily on Days 1 through 4 and a 30-mg daclatasvir tablet once daily along with an 800-mg darunavir tablet and a 100--mg ritonavir capsule once daily on Days 5 through 14.
Arm/Group | Group 1: Total | Group 1: Daclatasvir (60 mg) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir | Group 2: Total | Group 2: Daclatasvir (60 mg) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 6/14 | 1/14 | 6/14 | 8/14 | 3/14 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Total (N=14) | Group 1: Daclatasvir (60 mg) (N=14) | Group 1: Daclatasvir (30 mg) + Darunavir/Ritonavir (N=14) | Group 2: Total (N=14) | Group 2: Daclatasvir (60 mg) (N=14) | Group 2: Daclatasvir (30 mg) + Lopinavir/Ritonavir (N=14)
Electrocardiogram PR prolongation (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 5 | 0 | 5
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 1 | 3 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.